CLINICAL TRIAL: NCT04574362
Title: BHV3000-310: Phase 3: Double-Blind, Randomized, Placebo Controlled, Safety and Efficacy Trial of BHV3000 (Rimegepant) 75 mg for the Acute Treatment of Migraine
Brief Title: Safety and Efficacy Trial of BHV3000 (Rimegepant) 75 mg for the Acute Treatment of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: BioShin Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV3000-310; C4951026 (Other: Alias Study Number)
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-03

CONDITIONS: Acute Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rimegepant 75mg (Active Comparator): One 75mg oral disintegration tablet
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — One 75mg orally disintegrating tablet
  Arms: Rimegepant 75mg
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This trial is to determine whether BHV3000 (rimegepant) 75mg is safe and effictive as a treatment for acute migraine in Chinese and Korean patients

DETAILED DESCRIPTION:
Biohaven Pharmaceuticals, Inc. is the agent for BioShin Limited, the sponsor of the studies in China and Korea.

ELIGIBILITY:
Inclusion Criteria:

Subject has at least 1 year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorder, 3rd Edition, Beta version including the following:

1. Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age
2. Migraine attacks, on average, lasting about 4-72 hours if untreated
3. Not more than 8 attacks of moderate to severe intensity per month within the last 3 months
4. Consistent migraine headaches of at least 2 migraine headache attacks of moderate or severe intensity in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening period
5. Less than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening Period.
6. Subjects on prophylactic migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to screening visit and the dose is not expected to change during the course of the study.
7. Subjects with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Key Exclusion Criteria:

1. Subject with a history of HIV disease
2. Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. subjects with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening
3. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however subjects can be included who have stable hypertension and/or diabetes for at least 3 months prior to being enrolled)
4. Subject has a current diagnosis of major depression, other pain syndromes, psychiatric conditions (e.g., schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion might interfere with study assessments.
5. Subject has a history of gastric, or small intestinal surgery (including Gastric Bypass, Gastric Banding, Gastric Sleeve, Gastric Balloon, etc.), or has disease that causes malabsorption
6. The subject has a history of current or evidence of any significant and/ or unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial.
7. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months or subjects who have met DSM-V criteria for any significant substance use disorder within the past 12 months from the date of the screening visit.
8. Subjects are excluded if they have previously participated in any study of rimegepant or other experimental CGRP-antagonist study, or have been prescribed CGRP-antibodies within the last 6 months
9. Participation in any other investigational clinical trial while participating in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1648 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (90):
- China (77):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui provincal Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Lu'An People's Hospital, Lu'an, Anhui
  - The People's Hospital of Xuancheng City, Xuancheng, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Emergency Medical Center, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chonggang General Hospital, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Fujian medical University Union Hospital, Fuzhou, Fujian
  - The 900th Hospital of Joint Logistics Support Force, PLA, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Sun Yat-Sen Memorial Hospital of Zhongshan University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - Hainan General Hospital, Haikou, Hainan
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Henan University of Science and Technology First Affiliated Hospital, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huanggang Central Hospital, Huanggang, Hubei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Taihe Hospital, Shiyan, Hubei
  - Wuhan Fourth hospital, Wuhan, Hubei
  - Renmin Hospital Of Wuhan University, Wuhan, Hubei
  - Wuhan Third Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital Of Central South University, Changsha, Hunan
  - The Central Hospital of Shaoyang, Shaoyang, Hunan
  - The First People's Hospital of Yueyang, Yueyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Zigong First People's Hospital, Sichuan, Igong
  - The first affiliated hospital of Baotou medical college of Inner Mongolia university of science and technology, Baotou, Inner Mongolia
  - Affiliated Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital With Nanjing Medical University, Nanjing, Jiangsu
  - Sir Run Run Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi Integrated Traditional Chinese and Western Medicine Hospital, Wuxi, Jiangsu
  - Wuxi people's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - 1st Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - General Hospital of Ningxia Medical Hospital, Yinchuan, Ningxia
  - Baoji Central Hospital, Baoji, Shaanxi
  - Xi'an Gaoxin Hospital Co., Ltd, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People' Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Yan'an University Xianyang Hospital Co., Ltd, Xianyang, Shaanxi
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Nankai University, Tianjin Union Medical Center, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - The Fifth Affiliated Hospital of Xinjiang Medical University, Xinjiang, Uramqi
  - People's Hospital of Xinjiang Uygur Autonomous Region, Xinjiang, Wulumuqi
  - The Second Affiliated Hospital of Xinjiang Medical University, Xinjiang, Wulumuqi
  - The Second Affiliated hospital of Kunming Medical University, Kunming, Yunnan
  - Ruian People's Hospital, Rui’an, Zhejiang
- South Korea (13):
  - Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungnam National University Hospital, Daejeon
  - Nowon Eulji Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul

REFERENCES:
- [Derived] Yu S, Guo A, Wang Z, Liu J, Tan G, Yang Q, Zhang M, Yibulaiyin H, Chen H, Zhang Y, Croop R, Sun Y, Liu Y, Zhao Q, Lu Z. Rimegepant orally disintegrating tablet 75 mg for acute treatment of migraine in adults from China: a subgroup analysis of a double-blind, randomized, placebo-controlled, phase 3 clinical trial. J Headache Pain. 2024 Apr 16;25(1):57. doi: 10.1186/s10194-024-01731-4. PMID 38627638
- [Derived] Yu S, Kim BK, Guo A, Kim MH, Zhang M, Wang Z, Liu J, Moon HS, Tan G, Yang Q, McGrath D, Hanna M, Stock DA, Gao Y, Croop R, Lu Z. Safety and efficacy of rimegepant orally disintegrating tablet for the acute treatment of migraine in China and South Korea: a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2023 Jun;22(6):476-484. doi: 10.1016/S1474-4422(23)00126-6. PMID 37210098
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 1648 participants were enrolled and screened. A total of 217 participants were screen failures. Only 1431 participants were randomized. Out of 1431 participants, only 1342 participants were treated.
Pre-assignment Details: Participants were dispensed with 1 dose of study drug at randomization (baseline). Participants were required to administer pre-dispensed study drug only when the participants developed a migraine headache of moderate or severe intensity and completed all required migraine assessment questions in the electronic diary (eDiary), including their current most bothersome migraine symptom within 45 days of randomization.
Groups:
- Rimegepant 75 Milligram (mg): Participants were randomized to receive 1 orally disintegrating tablet of rimegepant 75 mg. Participants were followed up to 7 days post-dose.
- Placebo: Participants were randomized to receive placebo matched to rimegepant. Participants were followed up to 7 days post-dose.
Period: Overall Study
Arm/Group | Rimegepant 75 Milligram (mg) | Placebo
Started | 716 | 715
Treated | 668 | 674
Completed | 709 | 704
Not Completed | 7 | 11
Not completed — Other | 0 | 5
Not completed — COVID-19 | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Participant anxious to go to their hometown and withdrew from study | 1 | 0
Not completed — Participant refused to come to the hospital | 1 | 0
Not completed — Participant refused the visit | 1 | 0
Not completed — Participant quit early because of business trip | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all treated participants (all enrolled participants who took either of the study drug).
Groups:
- Rimegepant 75 mg: Participants were randomized to receive 1 orally disintegrating tablet of rimegepant 75 mg. Participants were followed up to for 7 days post-dose.
- Total: Total of all reporting groups
Arm/Group | Rimegepant 75 mg | Placebo | Total
Number analyzed (Participants) | 668 | 674 | 1342
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (10.13) | 37.7 (10.70) | 37.8 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 526 | 563 | 1089
  Male | 142 | 111 | 253
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Freedom From Pain at 2 Hours Post-dose
Description: Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (no pain) were considered to have freedom from pain. Exact 95 percent (%) confidence interval (CI) was based on Clopper-Pearson method.
Time Frame: 2 hours post-dose
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug, had a migraine of moderate or severe intensity at the time of treatment, and provided at least 1 post-treatment efficacy data point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants | 19.8 [16.9 to 23.1] | 10.7 [8.5 to 13.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.2, 95% CI 2-sided [5.4 to 13.0] — Risk difference and associated 95 percent (%) confidence interval (CI) were calculated from Mantel-Haenszel test, stratified by use of prophylactic medication and country. The risk difference was tested at a two-sided alpha level of 0.05

2. Primary Outcome: Percentage of Participants Who Had Freedom From Most Bothersome Symptoms (MBS) at 2 Hours Post-dose
Description: MBS included nausea, phonophobia or photophobia. MBS were measured using a binary scale as 0= absent, 1= present. Participants who had score of 0 (MBS absent) were considered to have freedom from MBS. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 2 hours post-dose
Population: mITT participants included all randomized participants who took study drug, had a migraine of moderate or severe intensity at the time of treatment, and provided at least 1 post-treatment efficacy data point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants | 50.5 [46.6 to 54.3] | 35.8 [32.1 to 39.5]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.8, 95% CI 2-sided [9.6 to 20.0] — Risk difference and associated 95% CI were calculated from Mantel-Haenszel test, stratified by use of prophylactic medication and country. The risk difference was tested at a two-sided alpha level of 0.05

3. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-dose
Description: Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants who reported a pain level of moderate or severe at baseline and then reported a pain level of none or mild at 2 hours post-dose, were considered to have pain relief. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 2 hours post-dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants | 66.5 [62.8 to 70.1] | 48.5 [44.7 to 52.4]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Within the family of key secondary endpoints, multiplicity was controlled using the Hochberg procedure; Risk Difference (RD) = 18.1, 95% CI 2-sided [13.0 to 23.3] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Who Functioned Normally at 2 Hours Post-dose
Description: Participants rated the level of disability they perceived as a result of their migraine in performing normal actions using following level of severity: normal function, mild impairment, severe impairment, or required bedrest. This outcome measure was analyzed only among those participants who reported any impairment at baseline. Percentage of participants with a response of "normal function" at the 2 hours post-dose were reported in this outcome measure.
Time Frame: 2 hours post-dose
Population: mITT participants included all randomized participants who took study drug, had a migraine of moderate or severe intensity at the time of treatment, and provided at least 1 post-treatment efficacy data point. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 545 | 551
Percentage of participants | 40.7 [36.6 to 45.0] | 23.8 [20.3 to 27.6]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Within the family of key secondary endpoints, multiplicity was controlled using the Hochberg procedure; Risk Difference (RD) = 16.9, 95% CI 2-sided [11.4 to 22.3] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Used Rescue Medication Within 24 Hours Post-dose
Description: Percentage of participants who used rescue medications within 24 hours of administration of study drug were reported in this outcome measure. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 24 hours post-dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants | 8.4 [6.4 to 10.8] | 20.0 [17.1 to 23.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Within the family of key secondary endpoints, multiplicity was controlled using the Hochberg procedure; Risk Difference (RD) = -11.5, 95% CI 2-sided [-15.0 to -8.0] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Sustained Pain Freedom From 2 to 24 Hours Post-dose
Description: Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (with no pain) through 2 to 24 hours post-dose were considered to have sustained pain freedom. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 2 to 24 hours post-dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants | 15.6 [12.9 to 18.6] | 7.9 [5.9 to 10.2]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Within the family of key secondary endpoints, multiplicity was controlled using the Hochberg procedure; Risk Difference (RD) = 7.7, 95% CI 2-sided [4.3 to 11.2] — Risk differences and associated 95% CI were calculated from Mantel-Haenszel test, stratified by use of prophylactic medication and country. The risk difference was tested at a two-sided alpha level of 0.05

7. Secondary Outcome: Percentage of Participants Who Sustained Pain Freedom From 2 to 48 Hours Post-dose
Description: Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (with no pain) through 2 to 48 hours post-dose were considered to have sustained pain freedom. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 2 to 48 hours post-dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants | 14.9 [12.2 to 17.8] | 7.1 [5.3 to 9.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Within the family of key secondary endpoints, multiplicity was controlled using the Hochberg procedure; Risk difference = 7.7, 95% CI 2-sided [4.4 to 11.0] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Percentage of Participants Who Had Freedom From Pain at 15, 30, 45, 60 and 90 Minutes Post-dose
Description: Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Percentage of participants who reported a pain level of moderate or severe just before taking study treatment and then reported a pain level of none at the specified timepoints. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 15, 30, 45, 60 and 90 minutes post-dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants
  15 minutes post-dose | 0.8 [0.2 to 1.7] | 1.5 [0.7 to 2.7]
  30 minutes post-dose | 1.1 [0.4 to 2.2] | 1.0 [0.4 to 2.1]
  45 minutes post-dose | 3.3 [2.1 to 5.0] | 2.2 [1.3 to 3.6]
  60 minutes post-dose | 6.8 [5.0 to 8.9] | 4.5 [3.0 to 6.3]
  90 minutes post-dose | 12.3 [9.9 to 15.1] | 7.1 [5.3 to 9.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; 15 minutes post-dose; Test type: Superiority; p = 0.2057, Cochran-Mantel-Haenszel — Nominal p-value; Risk difference = -0.7, 95% CI 2-sided [-1.9 to 0.4] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Rimegepant 75 mg vs Placebo; 30 minutes post-dose; Test type: Superiority; p = 0.9702, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 0.0, 95% CI 2-sided [-1.1 to 1.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Rimegepant 75 mg vs Placebo; 45 minutes post-dose; Test type: Superiority; p = 0.2419, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 1.0, 95% CI 2-sided [-0.7 to 2.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Rimegepant 75 mg vs Placebo; 60 minutes post-dose; Test type: Superiority; p = 0.0597, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 2.4, 95% CI 2-sided [-0.1 to 4.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Rimegepant 75 mg vs Placebo; 90 minutes post-dose; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 5.2, 95% CI 2-sided [2.1 to 8.4] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Percentage of Participants Who Had Freedom From MBS at 15, 30, 45, 60 and 90 Minutes Post-dose
Description: MBS included nausea, phonophobia or photophobia. MBS were measured using a binary scale as 0= absent, 1= present. Participants who had score of 0 (MBS absent) were considered to have freedom from MBS at the specified timepoints. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 15, 30, 45, 60 and 90 minutes post-dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 666 | 674
Percentage of participants
  15 minutes post-dose | 10.2 [8.0 to 12.8] | 11.1 [8.9 to 13.7]
  30 minutes post-dose | 16.8 [14.1 to 19.9] | 14.8 [12.2 to 17.7]
  45 minutes post-dose | 24.2 [21.0 to 27.6] | 19.9 [16.9 to 23.1]
  60 minutes post-dose | 31.1 [27.6 to 34.7] | 24.8 [21.6 to 28.2]
  90 minutes post-dose | 41.4 [37.7 to 45.3] | 31.8 [28.2 to 35.4]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; 15 minutes post-dose; Test type: Superiority; p = 0.6809, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = -0.7, 95% CI 2-sided [-3.9 to 2.5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Rimegepant 75 mg vs Placebo; 30 minutes post-dose; Test type: Superiority; p = 0.2586, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 2.2, 95% CI 2-sided [-1.6 to 6.0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Rimegepant 75 mg vs Placebo; 45 minutes post-dose; Test type: Superiority; p = 0.0421, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 4.5, 95% CI 2-sided [0.2 to 8.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Rimegepant 75 mg vs Placebo; 60 minutes post-dose; Test type: Superiority; p = 0.0066, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 6.6, 95% CI 2-sided [1.8 to 11.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Rimegepant 75 mg vs Placebo; 90 minutes post-dose; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = 9.9, 95% CI 2-sided [4.8 to 14.9] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Percentage of Participants With Pain Relapse
Description: Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. This outcome measure was analyzed only in those participants who were pain free at 2 hours post-dose. Percentage of participants who were pain free at 2 hours post-dose and then had a migraine of any pain severity (score 2 or 3 on the 4-point scale) within 48 hours after administration of study drug were considered to have pain relapse. Exact 95% CI was based on Clopper-Pearson method.
Time Frame: 2 Hours to 48 Hours Post-dose
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 132 | 72
Percentage of participants | 25.0 [17.9 to 33.3] | 33.3 [22.7 to 45.4]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.1148, Cochran-Mantel-Haenszel — Nominal p-value; Risk Difference (RD) = -10.4, 95% CI 2-sided [-23.5 to 2.8] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 7 days post-dose
Description: Same event may appear as adverse event and serious adverse event, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Treated population evaluated.
Arm/Group | Rimegepant 75 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/668 | 0/674
Serious Adverse Events (participants affected / at risk) | 1/668 | 2/674
Other Adverse Events (participants affected / at risk) | 92/668 | 94/674
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant 75 mg (N=668) | Placebo (N=674)
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Decreased embryo viability (Injury, poisoning and procedural complications) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant 75 mg (N=668) | Placebo (N=674)
Protein urine present (Investigations) | 8 | 7
Blood creatine phosphokinase increased (Investigations) | 5 | 3
Blood urine present (Investigations) | 3 | 2
Blood glucose increased (Investigations) | 3 | 1
Urine leukocyte esterase positive (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1
Urine ketone body present (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 0
Nitrite urine present (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 1
Urine analysis abnormal (Investigations) | 1 | 1
Weight increased (Investigations) | 2 | 0
White blood cells urine positive (Investigations) | 2 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatine phosphokinase MM increased (Investigations) | 0 | 1
Blood uric acid abnormal (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Crystal urine present (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 18
Vomiting (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Gingivitis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Erythropenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 3
Palpitations (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 4 | 1
Haematuria (Renal and urinary disorders) | 2 | 1
Albuminuria (Renal and urinary disorders) | 1 | 0
Photophobia (Eye disorders) | 4 | 3
Dizziness (Nervous system disorders) | 2 | 2
Burning sensation (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 2
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Phonophobia (Psychiatric disorders) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT04574362/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT04574362/SAP_001.pdf